CLINICAL TRIAL: NCT01601028
Title: Phase 3 Study of Hydroxychloroquine Treatment of Dry Eyes in Patients With Primary Sjögren's Syndrome
Brief Title: Hydroxychloroquine Treatment of Dry Eyes in Patients With Primary Sjögren's Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Hydroxychloroquine
Record Dates: First submitted 2012-04-29; First posted 2012-05-17 (Estimated); Last update posted 2013-10-17 (Estimated); Status verified 2013-10

CONDITIONS: Autoimmune Diseases; Sjogren's Syndrome; Dry Eye
Keywords: Autoimmune Diseases; Sjogren's Syndrome; Hydroxychloroquine
MeSH Terms: conditions — Autoimmune Diseases; Sjogren's Syndrome; Dry Eye Syndromes | interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hydroxychloroquine (Active Comparator): Hydroxychloroquine 300 mg once daily p.o.
  Interventions: Drug: Hydroxychloroquine
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine 300 mg once daily p.o. for 12 weeks and go off medication for 4 weeks (total 16 weeks)
  Arms: Hydroxychloroquine
Drug: Placebo — 2cp/day for 12 weeks and go off medication for 4 weeks (total 16 weeks)
  Arms: Placebo

SUMMARY:
Primary Sjögren syndrome is one of the most prevalent autoimmune diseases that present with dry eye and dry mouth. But there is no proven effective treatment for Sjögren syndrome patient. The relation between toll-like receptor (TLR) and the pathogenesis of Sjögren syndrome has been reported. Hydroxychloroquine is TLR7 and TLR9 antagonist. A few studies have been reported the effectiveness of Hydroxychloroquine for Sjögren syndrome but no randomized controlled study has been done. So the investigators evaluate the effectiveness and safeness of Hydroxychloroquine for primary Sjögren syndrome by randomized controlled study (Hydroxychloroquine 300 mg once daily p.o. group (N = 30) versus placebo group (N = 30).

ELIGIBILITY:
Inclusion Criteria:

* Patient who is diagnosed with primary Sjögren syndrome according to American/European consensus group (AECG) criteria
* Patient with the ability to give informed, dated and signed consent before the beginning of any proceedings related to the trial

Exclusion Criteria:

* Previous treated by Hydroxychloroquine but enough washout time after discontinuance of treatment, patient can be enrolled. (2 wks)
* Known cardiac disease, Respiratory disease, Renal disease, Gastrointestinal disease (except GERD)
* Diabetes mellitus
* Psoriasis
* Known drug allergy or hypersensitivity
* Previous or ongoing treatment by any drugs (include topical drug) which have effect on lacrimal system. But enough washout time after discontinuance of treatment, patient can be enrolled. (cf. SSRI, Anti-histamine, Pilocarpine, etc.)
* Angle closer glaucoma
* Patient who underwent previous intraocular surgery
* Macular disease
* Previous or ongoing treatment by drug which could have effect on macula
* Pregnancy
* Planning to get pregnant

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-07; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Serum cytokine level | 16 weeks
  IL-6, IL-17, IL-1b, TNF-alpha, INF-alpha, BAFF, etc.

SECONDARY OUTCOMES:
Retinal exam | 16 weeks
  Macular exam for monitoring Hydroxychloroquine macular toxicity
Indicator of inflammation | 16 weeks
  Serum ESR
Tear production | 16 weeks
  Schirmer's test
Subjective clinical eye complaints | 16 weeks
  Ocular Surface Disease Index (OSDI)
Tear cytokine level | 16 weeks
  IL-6, IL-17, IL-1b, TNF-alpha, INF-alpha, BAFF, etc.
Visual acuity | 16 weeks
  Best corrected visual acuity (Snellen)
Color test | 16 weeks
  HRR color vision test for monitoring hydroxychloroquine retinal toxicity
Tear breakup time | 16 weeks
  BUT (sec)
Corneal punctate fluorescein staining score | 16 weeks
  Corneal staining score (National Eye Institute Scale)
Changes in serum T-cell property | 16 weeks
  Serum T-cell property (FACS)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National Unversity Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Yoon CH, Lee HJ, Lee EY, Lee EB, Lee WW, Kim MK, Wee WR. Effect of Hydroxychloroquine Treatment on Dry Eyes in Subjects with Primary Sjogren's Syndrome: a Double-Blind Randomized Control Study. J Korean Med Sci. 2016 Jul;31(7):1127-35. doi: 10.3346/jkms.2016.31.7.1127. Epub 2016 Apr 20. PMID 27366013